CLINICAL TRIAL: NCT00121472
Title: The HeartMate II LVAS Pivotal Study Protocol, Bridge to Cardiac Transplantation
Brief Title: Thoratec HeartMate II Left Ventricular Assist System (LVAS) for Bridge to Cardiac Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC010230-1
Record Dates: First submitted 2005-07-12; First posted 2005-07-21 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure, Congestive; Ventricular Dysfunction; Cardiomyopathies
Keywords: Heart-assist devices
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Cardiomyopathies | interventions — Heart-Assist Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Thoratec HeartMate II Left Ventricular Assist System (LVAS) — Implantation of ventricular assist device to provide hemodynamic support
  Other Names: Thoratec; HeartMate II; Ventricular assist

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the Thoratec HeartMate II Left Ventricular Assist System (LVAS) as a bridge to cardiac transplantation in end-stage heart failure patients who are listed for cardiac transplant but are at imminent risk of dying.

The HeartMate II LVAS was approved by the US FDA on April 21, 2008, as a bridge to cardiac transplantation (reference PMA P060040). It was approved for commercial distribution in Canada on May 20, 2009 (reference Medical Device Licence #79765). Patients enrolled into the clinical trial will continue to be followed until all have reached a clinical outcome.

DETAILED DESCRIPTION:
The HeartMate II is a high speed, electric, axial flow, rotary blood pump. The pump drains blood from the left ventricular apex via a rigid inlet cannula and ejects into the aortic root via an outflow cannula joined to the aorta with an end to side anastomosis. Power and control of the pump are delivered through a percutaneous cable from the pump to the belt-worn System Driver. Patient outcomes will be compared to objective performance criteria based on historical data from other Thoratec implantable ventricular assist devices.

ELIGIBILITY:
Inclusion Criteria:

The following are general criteria; more specific conditions are included in the study protocol:

* Listed for cardiac transplantation
* NYHA Class IV heart failure symptoms
* On inotropic support, if tolerated
* Despite medical therapy, the patient must meet hemodynamic criteria for cardiogenic shock

Exclusion Criteria:

The following are general criteria; more specific conditions are included in the study protocol:

* Evidence of, or risk factors for end-organ dysfunction that would make LVAS implantation futile
* Existence of factors that would adversely affect patient survival or function of the LVAS.
* Intolerance to anticoagulant or antiplatelet therapies.
* Existence of any ongoing mechanical circulatory support other than intra-aortic balloon counterpulsation.
* Participation in any other clinical investigation that is likely to confound study results or affect study outcome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2005-03; Primary Completion 2006-11 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Thoratec Corporation
Locations (36):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Shands Hospital @ University of Florida, Gainesville, Florida
  - Methodist Hospital, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Barnes-Jewish Hospital/Washington University, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Columbia Presbyterian Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Hospital of University of PA, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Medical City Hospital Dallas, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin Medical School, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Hospital Royal Victoria / McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Result] Miller LW, Pagani FD, Russell SD, John R, Boyle AJ, Aaronson KD, Conte JV, Naka Y, Mancini D, Delgado RM, MacGillivray TE, Farrar DJ, Frazier OH; HeartMate II Clinical Investigators. Use of a continuous-flow device in patients awaiting heart transplantation. N Engl J Med. 2007 Aug 30;357(9):885-96. doi: 10.1056/NEJMoa067758. PMID 17761592
- [Derived] Brisco MA, Sundareswaran KS, Milano CA, Feldman D, Testani JM, Ewald GA, Slaughter MS, Farrar DJ, Goldberg LR; HeartMate II Clinical Investigators. Incidence, risk, and consequences of atrial arrhythmias in patients with continuous-flow left ventricular assist devices. J Card Surg. 2014 Jul;29(4):572-80. doi: 10.1111/jocs.12336. Epub 2014 Apr 18. PMID 24750460
- [Derived] Russell SD, Rogers JG, Milano CA, Dyke DB, Pagani FD, Aranda JM, Klodell CT Jr, Boyle AJ, John R, Chen L, Massey HT, Farrar DJ, Conte JV; HeartMate II Clinical Investigators. Renal and hepatic function improve in advanced heart failure patients during continuous-flow support with the HeartMate II left ventricular assist device. Circulation. 2009 Dec 8;120(23):2352-7. doi: 10.1161/CIRCULATIONAHA.108.814863. Epub 2009 Nov 23. PMID 19933938
- [Derived] Pagani FD, Miller LW, Russell SD, Aaronson KD, John R, Boyle AJ, Conte JV, Bogaev RC, MacGillivray TE, Naka Y, Mancini D, Massey HT, Chen L, Klodell CT, Aranda JM, Moazami N, Ewald GA, Farrar DJ, Frazier OH; HeartMate II Investigators. Extended mechanical circulatory support with a continuous-flow rotary left ventricular assist device. J Am Coll Cardiol. 2009 Jul 21;54(4):312-21. doi: 10.1016/j.jacc.2009.03.055. PMID 19608028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 486 patients were recruited at 36 cardiac transplantation hospitals between 8 Mar 2005 and 21 Apr 2008. After enrolling the initial 133 patients prespecified by the study protocol, an additional 353 patients were enrolled under a Continued Access Protocol(CAP) and in a concurrent Canadian study.
Pre-assignment Details: 194 patients were followed to at least 1 year after implantation of the device, all 133 of the Pivotal Study Cohort patients and 61 of the US CAP patients, results of which are summarized below and in the final FDA-approved labeling for the HeartMate II LVAS. The remaining 292 patients followed for less than 1 year are not included.
Groups:
- HeartMate II (HMII): HeartMate II Left Ventricular Assist System (HMII LVAS) used as a bridge to cardiac transplantation (133 Pivotal Study Cohort and 61 US Continued Access Protocol (CAP)).
Period: Overall Study
Arm/Group | HeartMate II (HMII)
Started | 194
Completed | 194 (Followed for at least 1 year after implantation of HM II LVAS.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HM II: HeartMate II LVAS used as a bridge to cardiac transplantation with at least 1-year follow-up (133 Pivotal Study Cohort and 61 US Continued Access Protocol)
Arm/Group | HM II
Number analyzed (Participants) | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 150
Body Surface Area [Mean (Standard Deviation); unit: sq. meter] — Body Surface Area (BSA) calculated from patients height and weight
  sq. meter | 1.99 (0.29)
Cardiac Index [Mean (Standard Deviation); unit: L/min/m^2] | 2.0 (0.5)
PCWP [Mean (Standard Deviation); unit: mmHg] — Pulmonary capillary wedge pressure
  mmHg | 26.0 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Survival to cardiac transplantation or 180 days on left ventricular assist system (LVAS) support while remaining listed for cardiac transplantation as United Network for Organ Sharing (UNOS)status 1A or 1B (please refer to www.unos.org for complete definitions of status).
Time Frame: 180 days
Population: The first consecutive 194 patients enrolled under the Pivotal Study Protocol (n=133) and the Continued Access Protocol (CAP, n=61) were analyzed when the last subject reached the 1 year followup point on September 14, 2007. Analysis was Intent To Treat (ITT).
Measure: Number; unit: participants
Groups:
- HM II: HeartMate II LVAS used as a bridge to cardiac transplantation (133 Pivotal Study Cohort and 61 US Continued Access Protocol (CAP).
Arm/Group | HM II
Number analyzed (Participants) | 194
participants
  Transplanted | 112
  Myocardial recovery, device removed | 6
  Alive on device at 180 days & UNOS Status 1A or 1B | 18
  Alive on device at 180 days, not Status 1A or 1B | 19
  Received other ventricular assist device | 3
  Expired prior to 180 days while on VAD support | 36

2. Secondary Outcome: Clinical Reliability (Malfunctions/Failures)
Description: Confirmed malfunctions/Serious Adverse Events
Time Frame: continuous
Measure: Number; unit: Number of Serious Events
Arm/Group | HM II
Number analyzed (Participants) | 194
Number of Serious Events
  Pump | 7
  Inflow Cannula | 2
  Outflow Cannula | 2
  System Controller | 10
  System Monitor | 0
  Display Module | 0
  Power Base Unit | 0
  Power Base Unit Cable | 1
  Batteries | 1
  Battery Clips | 0
  Shower Kit | 0
  Surgical Accessories | 0

3. Secondary Outcome: Kansas City Cardiomyopathy Questionaire (KCCQ)
Description: KCCQ is a validated instrument to self assess quality of life including physical function and social function. The instrument provides two scores, the Overall Summary (OSS) and Clinical Summary (CSS). Scores are calculated based on responses to the questionnaire, on a scale from 0-100. The higher the score, the better the quality of life. The patients' scores at six months were compared to their baseline scores and the resulting positive scores indicated improved quality of life.
Time Frame: baseline to 6 months
Population: Patients alive and capable of performing the test at 6 months
Measure: Mean (Standard Error); unit: Units on a KCCQ Score scale
Groups:
- HMII: HeartMate II LVAS used as a bridge to cardiac transplantation with at least 1-year follow-up (133 Pivotal Study Cohort and 61 US Continued Access Protocol)
Arm/Group | HMII
Number analyzed (Participants) | 53
Units on a KCCQ Score scale
  KCCQ Overall Summary Score (OSS) | 29.5 (2.7)
  KCCQ Clinical Summary Score (CSS) | 28.8 (2.4)

4. Secondary Outcome: New York Heart Association (NYHA) Classification
Description: NYHA relates symptoms to every day activities and patients quality of life. Class 1 = no limitations on physical activity Class 2 - slight limitation of physical activity Class 3 - marked limitation of physical activity Class 4 = unable to carry out any physical activity without discomfort
Time Frame: baseline, 1 month, 3 months, 6 months
Population: All patients who survived to interval are included.
Measure: Mean (Full Range); unit: units on NYHA scale
Arm/Group | HM II
Number analyzed (Participants) | 194
units on NYHA scale
  Baseline NYHA Class | 4.0 (0.1) [3 to 4]
  Month 1 NYHA Class | 2.2 (0.8) [1 to 4]
  Month 3 NYHA Class | 1.8 (0.7) [1 to 4]
  Month 6 NYHA Class | 1.7 (0.7) [1 to 3]

5. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire (MLWHF)
Description: MLWHF is a validated instrument to self assess how heart failure and its treatment affect the key physical, emotional, social and psychological dimensions of quality of life. The instrument is made up of 21 items that assess the patient's perception of these dimensions on a scale ranging from no (0) to very much (5). The total MLWHF score is calculated by adding the scores for all 21 items (range, 0-105). A lower score indicates a better quality of life. The patients' score at six months was compared to their baseline score and the resulting negative score indicates improved quality of life.
Time Frame: Baseline to 6 months
Population: Patients alive and capable of performing the test at 6 months
Measure: Mean (Standard Error); unit: units on a MLWHF Score scale
Groups:
- HMII: HeartMate II LVAS used as a bridge to cardiac transplantation (133 Pivotal Study Cohort and 61 US Continued Access Protocol (CAP).
Arm/Group | HMII
Number analyzed (Participants) | 52
units on a MLWHF Score scale | -32.3 (2.9)

6. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: The Six Minute Walk Test(6MWT)measures the distance that a patient can walk in a period of 6 minutes. The distance walked is measured in meters. This test measures the patients' functional status. The more meters a patient can walk over baseline indicates improvement in functional status.
Time Frame: baseline to 6 months
Population: Mean change from baseline in 6MWT distance at Month 1, 3, and 6. Only patients alive, capable and willing to perform test are included.
Measure: Mean (Standard Error); unit: meters
Arm/Group | HMII
Number analyzed (Participants) | 194
meters
  Month 1 (N = 151) | 149.2 (14.5)
  Month 3 (N = 101) | 235.4 (22.0)
  Month 6 (N = 64) | 296.8 (27.8)

7. Secondary Outcome: Reoperations
Description: Additional surgery after the initial implant operation
Time Frame: continuous
Population: as for outcome 1
Measure: Number; unit: Number of Events
Groups:
- HMII Replacement: HeartMate II LVAS used as a bridge to cardiac transplantation (133 Pivotal Study Cohort and 61 US Continued Access Protocol (CAP).
Arm/Group | HMII Replacement
Number analyzed (Participants) | 194
Number of Events
  HMII Replacement | 8
  Bleeding | 104
  Mediastinal exploration, evacuation and chest clos | 7
  Chest closure or reinforcement of closure | 32
  ICD placement or exchange | 8
  Evacuation of pericardial effusion | 1
  RVAD placemant or removal | 9
  Tracheostomy | 9
  Cholecystectomy, feeding tube placement, tracheost | 1
  Evacuation of pleural effusion, dialysis catheter | 1
  Feeding tube placement, chest tube placement | 1
  Left lower lobe wedge resection | 1
  LVAD evaluation and repair | 2
  Mediastinal exploration and evacuation | 1
  Mediastinal exploration , wound debridement, ICD r | 1
  Placement of chest tubes | 1
  Removal of foreign body | 1
  Total abdominal cholectomy with end-ileostomy | 1
  Device explant | 1
  Feeding tube placement | 1
  Mediastinal exploration, chest closure, gortex gra | 2
  Mediastinal exploration , evacuation, pacemaker re | 1
  Pericardial window | 1

8. Secondary Outcome: Post-transplant Survival
Description: 30 day and 1 year post transplant survival
Time Frame: 30 days, 1 year
Population: Patients (n=112) who recieved a cardiac transplant were followed at 30 day and 1 year post-transplant to determine if the device influenced post-transplant survival.
Measure: Number; unit: percentage of participants
Arm/Group | HM II
Number analyzed (Participants) | 112
percentage of participants
  Survival at 30 days (%) | 96
  Survival at 1 year (%) | 87

ADVERSE EVENTS:
Time Frame: From time of device implant to time of cardiac transplantation, permanent device removal, or death.
Description: Adverse events were documented by study site staff as they occured per protocol definitions. Adverse events were adjudicated by an independent Clinical Events Committee (CEC).
Arm/Group | HMII
Serious Adverse Events (participants affected / at risk) | 194/194
Other Adverse Events (participants affected / at risk) | 36/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HMII (N=194)
Bleeding (General disorders) | 117 (225)
Bleeding requiring surgery (Blood and lymphatic system disorders) | 56 (64)
Stroke (Nervous system disorders) | 17 (19)
Driveline infection (Infections and infestations) | 16 (20)
Pocket infection (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 35 (47)
Right heart failure (Cardiac disorders) | 36 (37)
Device thrombosis (Blood and lymphatic system disorders) | 3 (3)
Hemolysis (Blood and lymphatic system disorders) | 6 (6)
Other neurological (Nervous system disorders) | 15 (18) — Includes transient ischemic attachs (TIA) and non-stroke neurological events.
Local infection (Infections and infestations) | 45 (74)
Peripheral Thromboembolism (Blood and lymphatic system disorders) | 10 (11)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 53 (66)
Cardiac arrhythmias (Cardiac disorders) | 82 (135)
Renal failure (Renal and urinary disorders) | 25 (26)
Hepatic dysfunction (Hepatobiliary disorders) | 3 (3)
Psychological (Psychiatric disorders) | 3 (5)
Myocardial infarction (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HMII (N=194)
Bleeding (General disorders) | 16 (50) — Non-serious bleeding events
Localized Infection (General disorders) | 15 (44) — Non-serious localized infection
Driveline Infection (General disorders) | 10 (16) — Non-serious driveline infection
Cardiac Arrhythmias (General disorders) | 29 (69) — Non-serious cardiac arrhythmias
Psychological (General disorders) | 10 (10) — Non-serious psychological
Device Malfunctions (General disorders) | 36 (61) — Non-serious device malfunctions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No